CLINICAL TRIAL: NCT03074123
Title: Cortisol Response to Low Dose Cosyntropin Stimulation Test in the Late Afternoon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, leonard.saiegh, MD, Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0003-17BNZ
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Adrenal Insufficiency
Keywords: cosyntropin stimulation test; low-dose
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental): 20 healthy subjects will undergo low dose cosyntropin stimulation test. Serum and salivary cortisol will be measured just before cosyntropin administration and 30 minutes later.
  Interventions: Diagnostic Test: low-dose cosyntropin stimulation test

INTERVENTIONS:
Diagnostic Test: low-dose cosyntropin stimulation test — Each subject recruited in the study will undergo low dose cosyntropin stimulation test via intravenous short 2.5 cm plastic tube. 1 μg/ml ACTH aliquot stock solution will be pushed through, followed by 5 ml physiologic saline (0.9%). For each subject, serum and salivary cortisol will be measured just before cosyntropin administration and 30 minutes later.

SUMMARY:
Previous study showed that afternoon cosyntropin testing was associated with a sevenfold increased likelihood of failing the 1μg test. However, in that study, investigators used a 20.3 cm plastic tube, which might have led to uncompleted cosyntropin delivery. In ther current study investigators will study afternoon 1μg cosyntropin cortisol stimulation using a short 2.5 cm tube.

DETAILED DESCRIPTION:
In earlier studies investigators claimed that subnormal cortisol response using plastic tubes might result from cosyntropin adherence to the tube and loss of the delivered dosage. It was shown that 21.6-58.6% of ACTH dosage had not been recovered when pushed through 20.3 cm plastic tube, and loss of ACTH may be up to 70% when cosyntropin was delivered through a plastic 30 cm scalp vein set.

Moreover, it was previously shown that afternoon cosyntropin testing was associated with a sevenfold increased likelihood of failing the 1μg test. However, in that study, investigators used a 20.3 cm plastic tube, which might have led to uncompleted cosyntropin delivery. In ther current study investigators will study afternoon 1μg cosyntropin cortisol stimulation using a short 2.5 cm tube.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

Clinical suspicion of hypoadrenalism Medical condition or treatment that might alter blood cortisol levels Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Blood cortisol | one day
  Serum cortisol concentrations during intravenous low dose cosyntropin stimulation through short tube.

SECONDARY OUTCOMES:
Salivary free cortisol | one day
  Salivary free cortisol concentrations during intravenous low dose cosyntropin stimulation through short tube.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saiegh, Principal Investigator — Bni-Zion medical center
Locations (1):
- Mira Koch, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No